CLINICAL TRIAL: NCT05032521
Title: Treatment of Hyperlactatemia in Acute Circulatory Failure Based on Analysis of CO2: a Prospective Randomized Superiority Study (The LACTEL Study)
Acronym: LACTEL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GUINOT 2021-3
Record Dates: First submitted 2021-08-27; First posted 2021-09-02 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Hyperlactatemia; Actue Circulatory Failure
MeSH Terms: conditions — Hyperlactatemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard practice (Active Comparator)
  Interventions: Biological: collection of biological data; Other: collection of demographic, ventilatory, cardiac echocardiography, arterial and venous gas data; Procedure: Standard treatment
- algorithm (Experimental)
  Interventions: Biological: collection of biological data; Other: collection of demographic, ventilatory, cardiac echocardiography, arterial and venous gas data; Procedure: stratified treatment according to algorithm

INTERVENTIONS:
Biological: collection of biological data — collection of biological data
Other: collection of demographic, ventilatory, cardiac echocardiography, arterial and venous gas data — These data are usually measured continuously (monitoring of the resuscitation patient) and recorded on recorded on the resuscitation software.
Procedure: Standard treatment — usual management based on the use of drugs according to international recommendations
  Arms: standard practice
Procedure: stratified treatment according to algorithm — management based on arteriovenous CO2 gradient Stratification of drug use
  Arms: algorithm

SUMMARY:
The management of a patient with shock is based on improving tissue oxygenation through hemodynamic optimization. Lactate is a marker of tissue hypoperfusion commonly used in the ICU. In principle, hyperlactatemia can be caused by either increased tissue production (tissue hypoperfusion: type A), decreased lactate uptake (type B), or a combination of both mechanisms. It is important to correctly determine the cause(s) of hyperlactatemia, as this determines the treatment (expanders, inotrope, vasopressor, blood derivative transfusion), and the patient's morbidity and mortality. A classic example of this concept is volume expanders, which are frequently used to correct hyperlactatemia secondary to tissue hypoperfusion, but are associated with mortality if used excessively (fluid overload). In clinical practice, it is difficult to differentiate the exact causes of hyperlactatemia (type A and type B). From work carried out over the last 20 years in septic shock and then in other states of shock and in the operating theatre, it has been shown that the arteriovenous CO2 gradient (pCO2gap) measured from arterial and venous blood gases is a marker of tissue hypoperfusion with better predictive ability than the usual markers (clinical examination, SVO2....). Furthermore, when we relate pCO2gap to the arteriovenous O2 difference (pCO2gap /C(a-v)O2), this ratio allows us to distinguish with greater accuracy between states of acute circulatory failure associated with anaerobiosis (tissue hypoperfusion, type A) and those related to the underlying disease.

Also, several studies have demonstrated a strong ability of the pCO2gap and the pCO2gap/CavO2 ratio to predict the severity of shock, mortality of the shock patient, hyperlactatemia, and correction of hyperlactatemia with hemodynamic treatment. As a result, many authors have proposed algorithms for the management of shock patients based on the measurement of these CO2-derived indexes.

The hypothesis of this study is that the use of an algorithm based on CO2gap and the CO2gap/CavO2 ratio is superior in terms of correction of hyperlactatemia to usual practice based on clinical and macro-hemodynamics.

ELIGIBILITY:
Inclusion Criteria:

* Oral, free and informed consent obtained from a trusted person (health care proxy) or a close relative or consent in an emergency situation
* Adult patient managed in intensive care for whom the physician has decided on hemodynamic management because of signs of acute circulatory failure (systolic blood pressure < 90 mmHg, mean arterial pressure < 65 mmHg, or the need for infusion of vasopressors, skin mottling, diuresis < 0.5 mL/kg/h for a duration ≥ 2 hours, skin recoloring time > 3 sec
* Arterial lactate level ≥ 3 mmol L-1

Exclusion Criteria:

* Person not affiliated to national health insurance
* Person subject to a measure of legal protection (curatorship, guardianship)
* Person subject to limited judicial protection
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the number of patients with a lactate clearance of more than 10% (change of more than 10% between baseline and the level measured at 2 hours after management) at H2. | 2 hours after inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

REFERENCES:
- [Result] Guinot PG, Evezard C, Nguyen M, Pili-Floury S, Berthoud V, Besch G, Bouhemad B; Lactel Study Group. Treatment of Acute Circulatory Failure Based on Carbon Dioxide-Oxygen (CO2-O2) Derived Indices: The Lactel Randomized Multicenter Study. Chest. 2025 Apr;167(4):1068-1078. doi: 10.1016/j.chest.2024.11.021. Epub 2024 Nov 28. PMID 39615831
- [Derived] Caruso V, Besch G, Nguyen M, Pili-Floury S, Bouhemad B, Guinot PG; Lactel Study Group. Treatment of Hyperlactatemia in Acute Circulatory Failure Based on CO2-O2-Derived Indices: Study Protocol for a Prospective, Multicentric, Single, Blind, Randomized, Superiority Study (The LACTEL Study). Front Cardiovasc Med. 2022 Jun 23;9:898406. doi: 10.3389/fcvm.2022.898406. eCollection 2022. PMID 35811716